CLINICAL TRIAL: NCT02416531
Title: Vulvar Lichen Sclerosus: Therapeutic Comparison Between Clobetasol Propionate, Photodynamic Therapy and Low-Intensity Laser
Brief Title: Vulvar Lichen Sclerosus: Comparison Between Clobetasol Propionate, Photodynamic Therapy and Low-Intensity Laser
Acronym: VLSCBCPPTLIL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daniela de Fátima Teixeira da Silva (Other)
Collaborators: Hospital Perola Byington (Other Government)
Responsible Party: Sponsor-Investigator, Daniela de Fátima Teixeira da Silva, Professor of Postgraduate program in Biophotonics applied to HealthSciences, University of Nove de Julho
Organization: University of Nove de Julho (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Lichen-768168
Record Dates: First submitted 2015-03-25; First posted 2015-04-15 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Vulvar Lichen Sclerosus
Keywords: Vulvar lichen sclerosus; Photodynamic therapy; Low-level laser therapy; Clobetasol propionate
MeSH Terms: conditions — Vulvar Lichen Sclerosus | interventions — Clobetasol; Adrenal Cortex Hormones; Photochemotherapy; 1-phenyl-3,3-dimethyltriazene; Low-Level Light Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Corticosteroid (Active Comparator): Clobetasol propionate 0.05% ointment applied once daily at a dose of 1 g/application (1 g sachets) for 4 weeks.
  Interventions: Drug: Clobetasol propionate
- Photodynamic therapy (Experimental): Methylene blue 0.01% intralesional, λ = 660 ± 10 nm, P = 100 mW, PD = 510 mW/cm2, E = 4 J, ED = 20 J/cm2, t = 40 s, once a week for 4 weeks.
  Interventions: Radiation: Photodynamic therapy
- Low level laser therapy (Experimental): λ = 660 ± 10 nm, P = 100 mW, PD = 510 mW/cm2, E = 4 J, ED = 20 J/cm2, t = 40 s, once a week for 4 weeks.
  Interventions: Radiation: Low level laser therapy

INTERVENTIONS:
Drug: Clobetasol propionate — Clobetasol propionate 0.05% ointment applied once daily at a dose of 1 g/application (1 g sachets) for 4 weeks.
  Other Names: Corticosteroid
  Arms: Corticosteroid
Radiation: Photodynamic therapy — Methylene blue 0.01% intralesional, λ = 660 ± 10 nm, P = 100 mW, PD = 510 mW/cm2, E = 4 J, ED = 20 J/cm2, t = 40 s, once a week for 4 weeks
  Other Names: PDT
  Arms: Photodynamic therapy
Radiation: Low level laser therapy — λ = 660 ± 10 nm, P = 100 mW, PD = 510 mW/cm2, E = 4 J, ED = 20 J/cm2, t = 40 s, once a week for 4 weeks
  Other Names: LLLT
  Arms: Low level laser therapy

SUMMARY:
Vulvar lichen sclerosus (VLS) is a lymphocyte-mediated disease of unknown etiology that can cause intense itching as well stenosis, hindering the evacuation and urination. It can also limit the sex life due to severe local pruritus, pain and dyspareunia (pain during sexual intercourse). The standard treatment for this disease is the use of topical corticosteroids to reduce the clinical symptoms and to try to increase disease-free intervals. Photodynamic therapy (PDT), a treatment that associates a light radiation with a photosensitizing agent and low-level laser therapy (LLLT) are therapies that can promote effective immunomodulatory responses at the application site by means of photophysical and photochemical phenomena from the molecular to the systemic level, which promote their use in chronic dermatoses. The aim is to study and compare the effects of PDT, LLLT, and topical corticosteroid in VLS evaluating clinical, histological, immunohistochemical and spectroscopic responses. The study will be prospective, randomized, and controlled, in a population of 60 women with histological diagnoses of VLS, enrolled on the outpatient clinic of Genitoscopy Department of the Pérola Byington Hospital in São Paulo. There will be 3 treatments groups: PDT, LLLT and topical corticosteroid, where will be allocated by randomization 20 patients in each one. The clinical course will be monitored by measuring local temperature, itching, clamping (atrophy), and the appearance of the lesion. Histologically, the slides will be classified according to the Hewitt grading and will have the ordering of collagen fibers quantified. Immunohistochemical analysis will be done using the markers IFN-γ, TGF-β, CD4, CD8, IL-1, p53 and Ki-67. Finally, the spectroscopic evaluation will be done by reflectance. Descriptive and inferential statistical analyses will be conducted to compare the groups and for associations between different responses.

DETAILED DESCRIPTION:
Dosimetry and Experimental Groups: There is no dosimetric protocol established for the treatment of VLS with PDT, nor with LLLT. According to the literature, energy densities range from 9 to 150 J/cm2 and power densities from 40 to 700 mW/cm2, not to mention work that do not report the dosimetry used. As such, the dosimetry to be used in this study is based on a pilot clinical study performed by our group.

The patients will be randomized into 3 groups with 20 patients in each one:

Group GC: Corticosteroid over the whole vulva. Clobetasol propionate 0.05% ointment applied once daily at a dose of 1 g/application (1 g sachets) for 4 weeks.

Group GPDT: Localized photodynamic therapy at 8 points of the vulva. Methylene blue 0.01% intralesional, λ = 660 ± 10 nm, P = 100 mW, PD = 510 mW/cm2, E = 4 J, ED = 20 J/cm2, t = 40 s, once a week for 4 weeks.

Group GLLLT: Localized low-level laser therapy at 8 points of the vulva. The same parameters as for GPDT, except for the methylene blue, once a week for 4 weeks.

Analyses: The histological and immunohistochemical analyses will be performed before and 30 days after the start of treatment, whereas clinical analysis will be performed weekly on treatment days for the GPDT and GLLLT groups. The control group will not be seen weekly because the standard treatment is performed by the patients themselves, in their own homes, for 30 days as recommended by the International Society for the Study of Vulvar Disease (ISSVD).

After treatments the patients will be followed for verification of recorrence during one year, at minimum.

ELIGIBILITY:
Inclusion Criteria:

* adult female patients (aged over 18 years);
* vulvar lichen sclerosus diagnosed histologically;
* normal level of cortisol confirmed by blood test.

Exclusion Criteria:

* adult female patients under the age of 18;
* patients with any kind of ongoing cancer and/or AIDS or coagulopathy, pregnant or breastfeeding women;
* patients using corticosteroids, immunosuppressants or anticoagulants;
* patients with renal, hepatic or pulmonary-cardiovascular failure;
* patients who have undergone any kind of organ transplantation in the last three years.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in biopsies at 1 month. | Participants will be followed for 1 month during VLS's treatment.
  Biopsies will be performed at two points: at baseline to confirm the VLS and subsequent inclusion in the research protocol, and at the end of 30 days to investigate the prognosis after treatment.

SECONDARY OUTCOMES:
Count cells per mm2 by immunohistochemical reaction of IFN-γ, TGF-β, CD4, CD8, IL-1, p53 and Ki-67. | Participants will be followed for 1 month during VLS's treatment.
  Once deparaffinized, the tissue samples will be subjected to antigen retrieval, endogenous enzyme blocking, background blocking, incubations of antibodies, and counter-staining according to the instructions of the manufacturers. The cells that are positively stained by the immunohistochemical reaction will be counted with the aid of ImageJ software (National Institutes of Health, Maryland, USA) by two independent pathologists without prior knowledge of the experimental groups.
Percentage of relative reflectance as assessed by In-Vivo Reflectance Spectroscopy. | Participants will be followed for 1 month during VLS's treatment.
  A portable spectrophotometer (400-900 nm) comprising a light source and a fiber-optic probe will be used directly on the surface of the vulvar skin in areas affected by VLS and in healthy areas of the same patients. Relative spectra will be obtained for the wavelengths corresponding to those of the therapeutic window, and the percentage of relative reflectance will be calculated.
Temperature, as assessed by infrared thermographic camera, in Celsius degrees. | Participants will be followed for 1 month during VLS's treatment.
  Measurements will be recorded as images in all sessions before, during, and after irradiation to observe the thermal fluctuation in the procedures.
Itching, as assessed by Visual Analog Scale. | Participants will be followed for 1 month during VLS's treatment.
  In each session, the patients will be asked about the intensity of vulvar itching to assess its severity and duration, before and after irradiation, according to a visual analog scale.
Clamping, as assessed by digital caliper, in mm. | Participants will be followed for 1 month during VLS's treatment.
  The clamping of the lesion to monitor skin atrophy will be done before irradiation at each session, using a digital caliper, transversely and longitudinally in relation to the labia majora.
Area, as assessed by digital camera, in cm2. | Participants will be followed for 1 month during VLS's treatment.
  The appearance and area of the lesion will be monitored with a digital camera at every session, before irradiation. To facilitate measurements, a metric scale will be rested on all vulvas for the photos. The areas of the lesions will be quantified using ImageJ software (National Institutes of Health, Maryland, USA).
Collagen birefringence, as assessed by polarized light microscope, in nm. | Participants will be followed for 1 month during VLS's treatment.
  The correlation between birefringence and collagen ordering has been used since the 1960s. To the present date, polarized-light microscopy is an efficient method to quantify the change in collagen birefringence due to the effects of different agents. Since atrophy of the skin is a characteristic symptom of patients with VLS, the more detailed study of collagen fibers will elucidate the interaction of radiation with this type of tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Daniela FT Silva, PhD, Principal Investigator — University of Nove de Julho
Locations (1):
- Hospital Pérola Byington, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Kreuter A, Wischnewski J, Terras S, Altmeyer P, Stucker M, Gambichler T. Coexistence of lichen sclerosus and morphea: a retrospective analysis of 472 patients with localized scleroderma from a German tertiary referral center. J Am Acad Dermatol. 2012 Dec;67(6):1157-62. doi: 10.1016/j.jaad.2012.04.003. Epub 2012 Apr 24. PMID 22533994
- [Background] Oyama N, Chan I, Neill SM, Hamada T, South AP, Wessagowit V, Wojnarowska F, D'Cruz D, Hughes GJ, Black MM, McGrath JA. Autoantibodies to extracellular matrix protein 1 in lichen sclerosus. Lancet. 2003 Jul 12;362(9378):118-23. doi: 10.1016/S0140-6736(03)13863-9. PMID 12867112
- [Background] Gambichler T, Kammann S, Tigges C, Kobus S, Skrygan M, Meier JJ, Kohler CU, Scola N, Stucker M, Bechara FG, Altmeyer P, Kreuter A. Cell cycle regulation and proliferation in lichen sclerosus. Regul Pept. 2011 Apr 11;167(2-3):209-14. doi: 10.1016/j.regpep.2011.02.003. Epub 2011 Feb 15. PMID 21329728
- [Background] Terlou A, Santegoets LA, van der Meijden WI, Heijmans-Antonissen C, Swagemakers SM, van der Spek PJ, Ewing PC, van Beurden M, Helmerhorst TJ, Blok LJ. An autoimmune phenotype in vulvar lichen sclerosus and lichen planus: a Th1 response and high levels of microRNA-155. J Invest Dermatol. 2012 Mar;132(3 Pt 1):658-66. doi: 10.1038/jid.2011.369. Epub 2011 Nov 24. PMID 22113482
- [Background] Gambichler T, Terras S, Kreuter A, Skrygan M. Altered global methylation and hydroxymethylation status in vulvar lichen sclerosus: further support for epigenetic mechanisms. Br J Dermatol. 2014 Mar;170(3):687-93. doi: 10.1111/bjd.12702. PMID 24164308
- [Background] Perez-Lopez FR, Ceausu I, Depypere H, Erel CT, Lambrinoudaki I, Rees M, Schenck-Gustafsson K, Tremollieres F, van der Schouw YT, Simoncini T; EMAS, Spanish Menopause society. EMAS clinical guide: vulvar lichen sclerosus in peri and postmenopausal women. Maturitas. 2013 Mar;74(3):279-82. doi: 10.1016/j.maturitas.2012.12.006. Epub 2013 Jan 3. PMID 23291001
- [Background] Murphy R. Lichen sclerosus. Dermatol Clin. 2010 Oct;28(4):707-15. doi: 10.1016/j.det.2010.07.006. PMID 20883914
- [Background] Selim MA, Hoang MP. A histologic review of vulvar inflammatory dermatoses and intraepithelial neoplasm. Dermatol Clin. 2010 Oct;28(4):649-67. doi: 10.1016/j.det.2010.07.005. Epub 2010 Aug 30. PMID 20883910
- [Background] Monsalvez V, Rivera R, Vanaclocha F. [Lichen sclerosus]. Actas Dermosifiliogr. 2010 Jan-Feb;101(1):31-8. Spanish. PMID 20109390
- [Background] Brodrick B, Belkin ZR, Goldstein AT. Influence of treatments on prognosis for vulvar lichen sclerosus: facts and controversies. Clin Dermatol. 2013 Nov-Dec;31(6):780-6. doi: 10.1016/j.clindermatol.2013.05.017. PMID 24160287
- [Background] Hantschmann P, Sterzer S, Jeschke U, Friese K. P53 expression in vulvar carcinoma, vulvar intraepithelial neoplasia, squamous cell hyperplasia and lichen sclerosus. Anticancer Res. 2005 May-Jun;25(3A):1739-45. PMID 16033093
- [Background] Thorstensen KA, Birenbaum DL. Recognition and management of vulvar dermatologic conditions: lichen sclerosus, lichen planus, and lichen simplex chronicus. J Midwifery Womens Health. 2012 May-Jun;57(3):260-75. doi: 10.1111/j.1542-2011.2012.00175.x. PMID 22594865
- [Background] Lipkin D, Kwon Y. Therapies and nursing care of women with vulvar dermatologic disorders. J Obstet Gynecol Neonatal Nurs. 2014 Mar-Apr;43(2):246-52. doi: 10.1111/1552-6909.12286. Epub 2014 Feb 6. PMID 24502413
- [Background] Burrows LJ, Creasey A, Goldstein AT. The treatment of vulvar lichen sclerosus and female sexual dysfunction. J Sex Med. 2011 Jan;8(1):219-22. doi: 10.1111/j.1743-6109.2010.02077.x. Epub 2010 Oct 18. PMID 20955314
- [Background] Terras S, Gambichler T, Moritz RK, Stucker M, Kreuter A. UV-A1 phototherapy vs clobetasol propionate, 0.05%, in the treatment of vulvar lichen sclerosus: a randomized clinical trial. JAMA Dermatol. 2014 Jun;150(6):621-7. doi: 10.1001/jamadermatol.2013.7733. PMID 24696010
- [Background] Olejek A, Steplewska K, Gabriel A, Kozak-Darmas I, Jarek A, Kellas-Sleczka S, Bydlinski F, Sieron-Stoltny K, Horak S, Chelmicki A, Sieron A. Efficacy of photodynamic therapy in vulvar lichen sclerosus treatment based on immunohistochemical analysis of CD34, CD44, myelin basic protein, and Ki67 antibodies. Int J Gynecol Cancer. 2010 Jul;20(5):879-87. doi: 10.1111/IGC.0b013e3181d94f05. PMID 20606538
- [Background] Osiecka BJ, Nockowski P, Jurczyszyn K, Ziolkowski P. Photodynamic therapy of vulvar lichen sclerosus et atrophicus in a woman with hypothyreosis--case report. Photodiagnosis Photodyn Ther. 2012 Jun;9(2):186-8. doi: 10.1016/j.pdpdt.2012.02.002. Epub 2012 Mar 27. PMID 22594990
- [Background] Romero A, Hernandez-Nunez A, Cordoba-Guijarro S, Arias-Palomo D, Borbujo-Martinez J. Treatment of recalcitrant erosive vulvar lichen sclerosus with photodynamic therapy. J Am Acad Dermatol. 2007 Aug;57(2 Suppl):S46-7. doi: 10.1016/j.jaad.2006.04.005. No abstract available. PMID 17637374
- [Background] Hillemanns P, Untch M, Prove F, Baumgartner R, Hillemanns M, Korell M. Photodynamic therapy of vulvar lichen sclerosus with 5-aminolevulinic acid. Obstet Gynecol. 1999 Jan;93(1):71-4. doi: 10.1016/s0029-7844(98)00321-4. PMID 9916959
- [Background] Sotiriou E, Panagiotidou D, Ioannidis D. An open trial of 5-aminolevulinic acid photodynamic therapy for vulvar lichen sclerosus. Eur J Obstet Gynecol Reprod Biol. 2008 Dec;141(2):187-8. doi: 10.1016/j.ejogrb.2008.07.027. Epub 2008 Sep 7. No abstract available. PMID 18778886
- [Background] Biniszkiewicz T, Olejek A, Kozak-Darmas I, Sieron A. Therapeutic effects of 5-ALA-induced photodynamic therapy in vulvar lichen sclerosus. Photodiagnosis Photodyn Ther. 2005 Jun;2(2):157-60. doi: 10.1016/S1572-1000(05)00062-1. Epub 2005 Aug 3. PMID 25048675
- [Derived] Belotto RA, Chavantes MC, Tardivo JP, Euzebio Dos Santos R, Fernandes RCM, Horliana ACRT, Pavani C, Teixeira da Silva DF. Therapeutic comparison between treatments for Vulvar Lichen Sclerosus: study protocol of a randomized prospective and controlled trial. BMC Womens Health. 2017 Aug 10;17(1):61. doi: 10.1186/s12905-017-0414-y. PMID 28793884